CLINICAL TRIAL: NCT04110522
Title: Accelerating Psoriatic Arthritis Detection in Patients With Psoriasis: Direct-to-patient Administration of Screening Questionnaires (D2P Screening)
Brief Title: Psoriatic Arthritis D2P Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica Walsh (Other)
Responsible Party: Sponsor-Investigator, Jessica Walsh, Assistant Professor, Rheumatology, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB_00117215
Record Dates: First submitted 2019-09-13; First posted 2019-10-01 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriasis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention with Direct Access to Rheumatologist (Experimental): Psoriasis patients with no prior diagnosis of PsA randomized to receive intervention PsA questionnaire, including instructions on how to directly schedule a rheumatologic evaluation
  Interventions: Other: Direct to patient PsA Screening Questionnaire
- Intervention with Standard of Care Referral (Experimental): Psoriasis patients with no prior diagnosis of PsA randomized to receive intervention PsA questionnaire, including instructions to talk with their doctor about a referral to a rheumatologist
  Interventions: Other: Direct to patient PsA Screening Questionnaire
- Control (No Intervention): Psoriasis patients with no prior diagnosis of PsA randomized to not receive an intervention PsA questionnaire

INTERVENTIONS:
Other: Direct to patient PsA Screening Questionnaire — Patients randomized to an intervention group will be asked to complete and score the 5-item Psoriasis Epidemiology Screening Tool (PEST) questionnaire. Those patients with an elevated score (PEST ≥3 out of 5) will be advised to complete a rheumatologic evaluation for PsA.
  Arms: Intervention with Direct Access to Rheumatologist; Intervention with Standard of Care Referral

SUMMARY:
The overarching goal of this study is to develop a direct-to-patient screening approach that will improve early Psoriatic Arthritis (PsA) detection in patients with psoriasis. Previously developed screening questionnaires were intended for use in the setting of a doctor's office to assist providers with referral decisions. However, these screening questionnaires are infrequently used in routine practice because of limitations with time and resources. The study will aim to develop a practical screening strategy that does not require involvement from dermatologists (or other non-rheumatology providers) and can systematically reach a broad range of psoriasis patients, including patients not attending dermatology clinics. The researchers hypothesize that disseminating questionnaires directly to patients outside of a clinic setting (direct-to-patient approach) will educate patients about their PsA risk and improve early PsA diagnoses.

DETAILED DESCRIPTION:
Electronic medical record (EMR) systems will be used to identify psoriasis patients without a PsA diagnosis. Patients will be randomized to receive a PsA screening questionnaire (intervention group) or not receive a questionnaire (control group). Rates of rheumatologic evaluations and new PsA diagnoses will be compared between the groups, using EMRs to longitudinally track outcomes.

Intervention group patients who through the completion of the PsA Screening questionnaire positively self-screen for an elevated PsA risk will either be randomly invited to directly access a rheumatology appointment or instructed to talk with their doctor about a rheumatology referral. We will compare rates of rheumatologic evaluations and new PsA diagnoses between these groups to identify the best method for accessing rheumatology appointments.

To determine if PsA patients diagnosed after receiving a screening questionnaire differ from patients diagnosed via usual care; investigators will examine disease duration, severity, and comorbidities in patients receiving and not receiving the screening questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Have an International Classification of Diseases (ICD) code diagnosis of psoriasis but without a confirmed diagnosis of Psoriatic Arthritis prior to study initiation
* Be age 18 or older
* Be geographically located within a reasonable proximity to the Rheumatology study site

Exclusion Criteria:

* Have psoriasis and a confirmed diagnosis of psoriatic arthritis made or confirmed by a rheumatologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18000 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a new PsA diagnosis | 6 months
  The percentage of psoriasis patients with a new diagnosis of PsA will be compared between the Experimental Arms and the Control Arm, and compared between the two Experimental Arms (intervention with direct access to rheumatologist and intervention with standard of care referral)
Symptom duration | 6 months
  Average duration of baseline symptoms prior to PsA diagnosis in the Experimental Arms (intervention with direct access to rheumatologist and intervention with standard of care referral) will be compared to the average duration of baseline symptoms prior to PsA diagnosis in the Control Arm

SECONDARY OUTCOMES:
Percentage of patients who complete a rheumatologic evaluation | 6 months
  The percentage of psoriasis patients who complete a rheumatologic evaluation will be compared between the Experimental Arms and the Control Arm, and compared between the two Experimental Arms (intervention with direct access to rheumatologist and intervention with standard of care referral)
Time to initial PsA diagnosis after questionnaire dissemination | 6 months
  The average time to PsA diagnosis after dissemination of the questionnaire in the Intervention with Direct Access to Rheumatologist arm compared to the Intervention with Standard of Care Referral Arm
Time to rheumatologic evaluation after questionnaire dissemination | 6 months
  The average time to rheumatologic evaluation after dissemination of the questionnaire in the Intervention with Direct Access to Rheumatologist arm compared to the Intervention with Standard of Care Referral Arm
Severity of PsA Disability | 6 months
  Average work disability in PsA, as measured by the Work Productivity and Activity Impairment questionnaire score will be compared between the Experimental ams (intervention with direct access to rheumatologist and intervention with standard of care referral) and the Control Arm
Physical function level in PsA | 6 months
  Average physical function level in PsA, as measured by the Health Assessment Questionnaire Disability Index (HAQ-DI) questionnaire score will be compared between the Experimental Arms (intervention with direct access to rheumatologist and intervention with standard of care referral) and the Control Arm.
Severity of PsA radiographic damage | 6 months
  Average number of psoriatic arthritis inflammatory changes per rheumatology provider's judgement after review of all relevant available imaging data using scale of yes/no/unsure will be compared between the Experimental Arms (intervention with direct access to rheumatologist and intervention with standard of care referral) and the Control Arm.
PsA Activity by Joint Count | 6 months
  Average number of swollen/tender joints in PsA using the 66/68 joint count assessment by rheumatology provider physical exam will be compared between the Experimental Arms (intervention with direct access to rheumatologist and intervention with standard of care referral) and the Control Arm.
PsA Activity by Enthesitis | 6 months
  Average number of joint insertions with enthesitis in PsA as determined by the Leeds enthesitis index as assessed by rheumatology provider physical exam will be compared between the Experimental Arms (intervention with direct access to rheumatologist and intervention with standard of care referral) and the Control Arm.
PsA Activity by Dactilitis Count | 6 months
  Average number of digits with dactylitis in PsA using a dactylitis count (yes/no for each finger or toe) as assessed by rheumatology provider physical exam will be compared between the Experimental Arms (intervention with direct access to rheumatologist and intervention with standard of care referral) and the Control Arm.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Walsh, M.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No